CLINICAL TRIAL: NCT06266247
Title: Relationship of Inflammation Markers and Sirtuin Levels Disease Activity in Patients With Behcet's Disease
Brief Title: How Sirtuin Levels Change During Behçet Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hilal Ecesoy, MD, Clinical profesor, Karamanoğlu Mehmetbey University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 06-2023/16; KMU-BAP (Other: KMU)
Record Dates: First submitted 2024-01-25; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Behçet Disease; Inflammation; Vasculitis
Keywords: Behçet; inflammation
MeSH Terms: conditions — Behcet Syndrome; Inflammation; Vasculitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Other): 1. Group: Behcet patients
  2. Group: Healty people
  Interventions: Diagnostic Test: Take blood samples

INTERVENTIONS:
Diagnostic Test: Take blood samples — Tnf alpha, sirtuin and il-6 levels will be examined in patients with Behcet's disease using biological drugs and not using biological drugs

SUMMARY:
Our primary aim in our study is to evaluate the relationship between the activity, which will be evaluated by clinical and standard phase reactants, and the IL-6 and TNF-α levels, which will be measured in serum, in Behçet's patients. Our secondary aim was to evaluate Sirtuin-1 in Behcet's patients and compare it with the normal population. Our third aim is to find out whether there is a relationship between these values and organ involvement.

DETAILED DESCRIPTION:
Behçet's disease (BD) is a systemic disease that has a long-term course with attacks, can involve many organs, and whose main pathology is vasculitis. For the first time in 1937 It was defined by Prof. Dr. Hulusi Behçet as a three-symptom complex consisting of hypopyonous uveitis along with oral and genital ulcers.

In recent years, especially as a result of developments in molecular biology, new information obtained about the structure and functions of immune system elements has revealed that the immune system plays an important role in the onset or course of the disease. Cytokines [such as IL-2, IL-6, IL-8, IL-12, Tumor Necrosis Factor-alpha (TNF-α) and Interferongama (IFN-γ)produced by Th-1 lymphocytes] that play important roles in inflammation in BD. It has been reported that the level of proinflammatory cytokines increases especially during the active period of the disease. It has been suggested that these cytokines may cause acute inflammatory tissue damage by causing neutrophil activation.

Sirtuins are known to be from the protein deacetylase and adenosine diphosphate (ADP)-ribosyl transferase protein families. Seven Sirtuin types have been identified in mammals (SIRT 1-7). Mammalian sirtuins can be affected in many physiological events such as metabolism, aging, cancer, and inflammation. Sirtuin 1 (SIRT1), a nicotinamide adenine dinucleotide (NAD+)-dependent histone deacetylase, has been reported to participate in the regulation of various biological processes such as energy balance, inflammation, oxidative stress, and mitochondrial biogenesis.

Our aim here is to compare cytokine levels according to organ involvement, drug used and to evaluate disease progression.

Blood samples for serum for cytokines and plasma for sirtuin will be taken from patients diagnosed with Behçet's disease between the ages of 18-65 who come to the Rheumatology Polyclinic for their normal routine check-up. The obtained samples will be stored at -80 °C until the blood of all patients is collected. In the control group, blood will be taken on a voluntary basis from people of appropriate age and gender who come to the polyclinic and do not have any inflammatory disease, and from hospital staff who do not have any health problems and do not use any medication.

All patients' name, surname, age, gender, family history of Behçet's disease, smoking-alcohol use, height-weight, additional diseases and medications used for Behçet's disease will be questioned. Blood pressure measurement, detailed physical and dermatological examination will be performed. Behçet's patients will be questioned in terms of oral aphthous ulcers, genital ulcers, erythema nodosum-like lesions, papulopustular lesions, arthritis, arthralgia, uveitis, vascular involvement, neurological involvement and gastrointestinal involvement.

The disease activity of Behçet patients at the time of admission will be determined using the Behçet Disease activity form.

Descriptive statistical methods (mean, standard deviation, median, frequency, ratio, minimum, maximum) will be used when evaluating study data. The suitability of quantitative data for normal distribution will be tested with the Kolmogorov-Smirnov and Shapiro-Wilk tests. Independent t Test will be used for two-group comparisons of normally distributed quantitative data, and Mann Whitney U test will be used for two-group comparisons of non-normally distributed data. One-way Anova Test was used for comparisons of three or more normally distributed groups, and Bonferroni test was used for pairwise comparisons. The Kruskal Wallis test will be used for comparisons of three or more groups that do not show normal distribution, and the Bonferroni-Dunn test will be used for pairwise comparisons. Pearson Chi-Square Test and Fisher's Exact Test will be used in comparisons of qualitative data. Spearman's Correlation Analysis will be used to evaluate the relationships between quantitative variables. Significance will be evaluated at at least p<0.05. (SPSS) program will be used for the evaluation

ELIGIBILITY:
Inclusion Criteria:

• Patients diagnosed with Behçet's disease between the ages of 18-65 who come to the Rheumatology Polyclinic for their normal routine check-up.

Exclusion Criteria:

* Suffer from other arthritis or joint diseases;
* Combined with severe liver and kidney function damage or metabolic diseases (such as thyroid and parathyroid diseases), affecting bone metabolism;
* Combined with serious cardiovascular and cerebrovascular diseases or chronic kidney diseases;
* Combined with tumour and bone metastasis;
* Taking anticancer drugs or other drugs that affect bone metabolism;
* Pregnant or lactating women;
* Exclude other autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Our primary aim is to evaluate the relationship between the activity to be evaluated with clinical and standard acute phase reactants and the IL-6 and TNF-α levels to be measured in serum in Behçet's patients. | From enrollment to the end of treatment at 6 months"
  Since Behçet's disease is an inflammatory disease, immediate blood samples will be taken from patients presenting to the outpatient clinic. Acute phase reactants, tnf-alpha levels and interleukin-6 levels will be measured. Behçet's disease current activity form 2006 (BDCAF-2006) will be filled and disease activity levels will be evaluated. BDCAF-2006 and acute phase reactants, tnf-alpha levels and interleukin-6 levels will be compared. The same comparison will be made with acute phase reactants, tnf-alpha levels and interleukin-6 levels in the blood obtained from the control group. The difference between both groups will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoğlu Mehmetbey University, Karaman, Turkey (Türkiye)